CLINICAL TRIAL: NCT01427686
Title: Effect of Dobutamine as Compared to Dopamine on Cerebral Oxygenation, Mean Arterial Pressure and Cerebral Hemodynamics in Term and Preterm Neonates With Arterial Hypotension
Brief Title: Dopamine Versus Dobutamine for Treatment of Arterial Hypotension in Term and Preterm Neonates
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manuel Schmid, Dr. med., University of Ulm
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ULMNEONIRS01
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Arterial Hypotension
MeSH Terms: conditions — Hypotension | interventions — Dobutamine; Dopamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dobutamine (Active Comparator): Start Dobutamine. If no success switch to Dopamine.
  Interventions: Drug: Dobutamine
- Dopamine (Active Comparator): Start Dopamine. If no success switch to Dobutamine.
  Interventions: Drug: Dopamine

INTERVENTIONS:
Drug: Dobutamine — Start Dobutamine with 5µg/kg/min. Increase as needed until mean arterial pressure is in normal range (defined by responsible neonatologist, usually between gestational age in weeks and 10mmHg above this threshold) or until a maximum dose of 15µg/kg/min is reached. Only in the latter case switch to Dopamine.
  Arms: Dobutamine
Drug: Dopamine — Start Dopamine with 5µg/kg/min. Increase as needed until mean arterial pressure is in normal range (defined by responsible neonatologist, usually between gestational age in weeks and 10mmHg above this threshold) or until a maximum dose of 15µg/kg/min is reached. Only in the latter case switch to Dobutamine.
  Arms: Dopamine

SUMMARY:
The purpose of this study is to examine the effects of Dobutamine as compared to Dopamine in term and preterm neonates with arterial hypotension on cerebral and renal oxygenation, fractional tissue oxygen extraction, mean arterial blood pressure and cardiac output.

The investigators hypothesize that Dopamine has a stronger effect on blood pressure than Dobutamine but Dobutamine has a stronger effect on cerebral oxygenation and cardiac output than Dopamine.

ELIGIBILITY:
Inclusion Criteria:

* fluid refractory arterial hypotension
* newborn infant below 44 weeks postmenstrual age
* parental informed consent

Exclusion Criteria:

* preterm infant below 28 weeks postmenstrual age during the first week of life
* congenital life-threatening malformations
* decision for palliative care
* hemorrhagic shock
* other obvious cause for arterial hypotension that requires immediate specific treatment, e.g. tension pneumothorax

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-02 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral tissue oxygen saturation | during study medication
  Cerebral tissue oxygen saturation (and derived parameters FTOE, HbD and Total Hb as secondary outcomes) measured by near-infrared spectroscopy after achieving normal blood pressure

SECONDARY OUTCOMES:
Cardiac output | during treatment
  Cardiac output and derived parameters (Cardiac index, stroke volumen, stroke index) as measured by electrical cardiovelocimetry
Cardiac output | during study medication
  Cardiac output and derived parameters (Cardiac index, stroke volumen, stroke index) as measured by electrical cardiovelocimetry

CONTACTS AND LOCATIONS:
Overall Officials: Manuel B Schmid, Dr. med., Principal Investigator — University of Ulm
Locations (1):
- University Medical Center, Ulm University, Ulm, Baden-Wurttemberg, Germany